CLINICAL TRIAL: NCT03737435
Title: Tumor Microenvironment in Patients With Localized Osteosarcoma Treated With Mifamurtide: a Translational Study
Acronym: Micros
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Micros
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Localized Osteosarcoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — archival samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
International, multicenter retrospecitve biological study

DETAILED DESCRIPTION:
International, multicenter retrospecitve biological study that will analyze the tumor micro environment in biological archival samples of patients, who were treated with chemotherapy +/- mifamurtide according the protocols for primary localized osteosarcoma (ISG-OS2 and GEIS-33)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary localized osteosarcoma who received chemotherapy +/- mifamurtide according to ISG-OS2/GEIS-33 trials,
2. Paraffin-embedded tissue tumor (FFPE) blocks from archive available to perform the biological analysis
3. Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

1) Patients with diagnosis different from osteosarcoma

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: male and female without limit of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Characterize the immunephenotype in patients with localized osteosarcoma treated with chemotherapy +/- mifamurtide for primary osteosarcoma | at baseline (Day0)
  A gene expression profile analysis will be performed through NanoString, using the PanCancer Immune Profiling Panel, which includes 770 genes related to the tumor microenvironment. This analysis will be carried out on the NanoString platform, present at the Hemolympopathology Division of the European Institute of Oncology
Correlate the rate of immune cells, and the level of the PDL-1 checkpoint with event-free survival and overall-survival | at baseline (Day0)
  For survival analysis the following factors will be correlated with Overall Suvival and Event Free Survival age (pediatric < 18 years vs adult ≥ 18 years), gender, LDH and phosphatase alkaline (PA) levels at baseline (normal vs high), pathologic response (good: chemotherapy-induced tumor necrosis ≥ 90%; poor: chemotherapy-induced tumor necrosis < 90%, [10]), tumoral miroenvironment components, PD-1 expression on IC, and PD-L1 both on TC and IC., genetic signatures.

CONTACTS AND LOCATIONS:
Locations (1):
- SSD Chemioterapia dei tumori dell'apparato locomotore, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palmerini E, Agostinelli C, Picci P, Pileri S, Marafioti T, Lollini PL, Scotlandi K, Longhi A, Benassi MS, Ferrari S. Tumoral immune-infiltrate (IF), PD-L1 expression and role of CD8/TIA-1 lymphocytes in localized osteosarcoma patients treated within protocol ISG-OS1. Oncotarget. 2017 Dec 4;8(67):111836-111846. doi: 10.18632/oncotarget.22912. eCollection 2017 Dec 19. PMID 29340095
- [Result] Koirala P, Roth ME, Gill J, Piperdi S, Chinai JM, Geller DS, Hoang BH, Park A, Fremed MA, Zang X, Gorlick R. Immune infiltration and PD-L1 expression in the tumor microenvironment are prognostic in osteosarcoma. Sci Rep. 2016 Jul 26;6:30093. doi: 10.1038/srep30093. PMID 27456063
- [Result] Dumars C, Ngyuen JM, Gaultier A, Lanel R, Corradini N, Gouin F, Heymann D, Heymann MF. Dysregulation of macrophage polarization is associated with the metastatic process in osteosarcoma. Oncotarget. 2016 Nov 29;7(48):78343-78354. doi: 10.18632/oncotarget.13055. PMID 27823976
- [Result] Picci P, Bacci G, Campanacci M, Gasparini M, Pilotti S, Cerasoli S, Bertoni F, Guerra A, Capanna R, Albisinni U, et al. Histologic evaluation of necrosis in osteosarcoma induced by chemotherapy. Regional mapping of viable and nonviable tumor. Cancer. 1985 Oct 1;56(7):1515-21. doi: 10.1002/1097-0142(19851001)56:73.0.co;2-6. PMID 3861228
- [Result] Meyers PA, Schwartz CL, Krailo M, Kleinerman ES, Betcher D, Bernstein ML, Conrad E, Ferguson W, Gebhardt M, Goorin AM, Harris MB, Healey J, Huvos A, Link M, Montebello J, Nadel H, Nieder M, Sato J, Siegal G, Weiner M, Wells R, Wold L, Womer R, Grier H. Osteosarcoma: a randomized, prospective trial of the addition of ifosfamide and/or muramyl tripeptide to cisplatin, doxorubicin, and high-dose methotrexate. J Clin Oncol. 2005 Mar 20;23(9):2004-11. doi: 10.1200/JCO.2005.06.031. PMID 15774791

DOCUMENTS (1):
  • Study Protocol (2020-02-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT03737435/Prot_001.pdf